CLINICAL TRIAL: NCT06157775
Title: Reliability of Ultrasound Shear-wave Elastography in Assessing Tensor Fascia Lata, Gluteus Medius, and Iliotibial Band Elasticity in Health Individuals: a Cross-sectional Study.
Brief Title: Shear-wave Elastography of Hip Stabilizers in Healthy Individuals
Status: Completed | Type: Observational
Sponsor: Koç University (Other)
Responsible Party: Sponsor
Other Study IDs: 2019.347.IRB1.062
Record Dates: First submitted 2023-11-20; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2019-10

CONDITIONS: Shear-wave Elastography of Hip Stabilizers in Healthy Individuals

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Healthy Individuals
  Interventions: Diagnostic Test: Shear-wave elastography

INTERVENTIONS:
Diagnostic Test: Shear-wave elastography — Shear-wave elastography using a manual ultrasound with a 9L-Probe in B-mode.

SUMMARY:
The aim of this study is to provide a scientific basis for Shear-wave elastography measurements of hip stabilizing muscles on healthy individuals. To assess the inter- and intra-user validity, 12 healthy volunteers were recruited for ultrasonographic assessment by two experienced physiatrists.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Individuals
* Age 18-30 years
* Volunteering for the study
* Absence of musculoskeletal pathologies involving pelvic, hip, and/or knee joints.

Exclusion Criteria:

* Recent complaints of pelvic, hip, and/or knee pain.
* Previous history of trauma or surgery, including the lumbar, pelvic, hip, or knee region.
* Congenital or acquired pathologies of pelvis or lower extremity.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 12 Healthy Individuals, 4 male and 8 female.
Sampling Method: Non-Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-10-31 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
Assessment of tensor fascia latae muscle on shear wave elastography. | 1 month
Assessment of gluteus medius muscle on shear wave elastography. | 1 month
Assessment of iliotibial band on shear wave elastography. | 1 month

CONTACTS AND LOCATIONS:
Overall Officials: Ozden Ozyemisci Taskiran, MD, Principal Investigator — Koc University Hospital
Locations (1):
- Koc University School of Medicine, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cortez CD, Hermitte L, Ramain A, Mesmann C, Lefort T, Pialat JB. Ultrasound shear wave velocity in skeletal muscle: A reproducibility study. Diagn Interv Imaging. 2016 Jan;97(1):71-9. doi: 10.1016/j.diii.2015.05.010. Epub 2015 Jun 25. PMID 26119864
- [Background] Iida N, Kuroiwa T, Amadio P. Analysis of the thenar muscles with ultrasound shear wave elastography: Reliability and preliminary findings. Muscle Nerve. 2024 Jan;69(1):72-77. doi: 10.1002/mus.28004. Epub 2023 Nov 15. PMID 37964671
- [Background] Whittaker JL, Emery CA. Sonographic measures of the gluteus medius, gluteus minimus, and vastus medialis muscles. J Orthop Sports Phys Ther. 2014 Aug;44(8):627-32. doi: 10.2519/jospt.2014.5315. Epub 2014 Jul 16. PMID 25029916
- [Background] Vuorenmaa AS, Siitama EMK, Makela KS. Inter-operator and inter-device reproducibility of shear wave elastography in healthy muscle tissues. J Appl Clin Med Phys. 2022 Sep;23(9):e13717. doi: 10.1002/acm2.13717. Epub 2022 Jul 6. PMID 35793227
- [Background] Gyaran IA, Spiezia F, Hudson Z, Maffulli N. Sonographic measurement of iliotibial band thickness: an observational study in healthy adult volunteers. Knee Surg Sports Traumatol Arthrosc. 2011 Mar;19(3):458-61. doi: 10.1007/s00167-010-1269-z. Epub 2010 Oct 2. PMID 20890700